CLINICAL TRIAL: NCT04538469
Title: Absent Visitors: The Wider Implications of COVID-19 on Non-COVID Cardiothoracic ICU Patients, Relatives and Staff
Acronym: VINCI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Glasgow (Other)
Collaborators: Golden Jubilee National Hospital (Other Government)
Responsible Party: Principal Investigator, Dr Ben Shelley, Chief Investigator, University of Glasgow
Other Study IDs: 20/ANAES/02
Record Dates: First submitted 2020-09-01; First posted 2020-09-04 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Cardiovascular Diseases; Delirium; Critical Illness; Intensive Care Unit Delirium; Thoracic Diseases; Respiratory Failure; Cardiac Disease; Cardiac Failure
MeSH Terms: conditions — Cardiovascular Diseases; Delirium; Critical Illness; Thoracic Diseases; Respiratory Insufficiency; Heart Diseases; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Admitted prior to COVID visitation restrictions introduced
- Group 2: Admitted following the introductions of visitation restrictions due to COVID 19 pandemic
  Interventions: Other: COVID visitation restrictions

INTERVENTIONS:
Other: COVID visitation restrictions — Visitation to patients in hospitals in Scotland was ceased due to the COVID 19 pandemic. Slow reintroduction of visitors has been introduced, however not to the pre COVID 19 levels. This study will examine the effects of these restrictions on patients in the cardiothoracic critical care unit that do not suffer from COVID 19.
  Groups: Group 2

SUMMARY:
Patients are part of a family network. When any person in a family becomes critically unwell and requires the assistance of an Intensive Care Unit (ICU), this has an impact on all members of that family.

COVID-19 changed visiting for all patients in hospitals across Scotland. It is not known what effect these restrictions will have on patients' recovery, nor do we understand the impact it may have on their relatives or staff caring for them. This study will look at the implications of the visiting restrictions as a consequence of the COVID-19 pandemic upon patients without COVID-19 who are in the cardiothoracic ICU. It will also explore the impact of these restrictions on them, their relatives and staff.

This study will be carried out within a single specialised intensive care unit in Scotland using mixed methods.

The first arm of this study will use retrospective data that is routinely collected in normal clinical practice. The investigators will compare patient outcomes prior to COVID-19 with outcomes following the implementation of COVID-19 visiting restrictions. The aim is to establish if the restrictions on visiting has an impact on the duration of delirium. Delirium is an acute mental confusion and is associated with longer hospital stays and worse outcomes in this patient group.

The second arm of this study involves semi-structured interviews with patients, relatives and staff that will allow deeper exploration of the issues around current visiting policy. The interviews will last approximately 1 hour and will address these issues. They will then be transcribed word for word and analysed using grounded theory, meaning the theories will develop from the data as it is analysed.

DETAILED DESCRIPTION:
This study will look at the implications of visiting restrictions on patients without COVID-19 who are in the intensive care unit. It will also explore the impact of these restrictions on them, their relatives and staff.

The investigators hypothesise that the restriction of visiting has a negative impact on recovery of patients, families of patients and staff caring for patients without COVID-19 in the cardiothoracic ICU.

In order to answer this hypothesis, the wider implications of COVID-19 will be explored, not only with patients, but also relatives and staff involved in the care of these patients.

The research questions this study aims to answer are:

1. Is there a negative impact on the clinical outcomes due to the COVID-19 visitation restrictions?
2. Is there an increase in the incidence and duration of delirium in patients who do not receive visitors?
3. What experiences do patients recall during their ICU admission through the COVID-19 pandemic visitation restrictions?
4. What experiences do relatives recall from their loved-ones during an ICU admission during the COVID-19 pandemic visitation restrictions?
5. What impact, if any, do the changes to visiting have on staff?

In order to answer these research questions the investigators will carry out a single centre mixed method observational study. This study will consist of two arms.

The first arm of this study will utilise retrospective data that is routinely collected in normal clinical practice in this single centre. This will be used to compare to patient outcomes prior to COVID-19 with outcomes following the implementation of COVID-19 visiting restrictions.

The second arm of this study involves semi-structured interviews with patients, relatives and staff that allow deeper exploration of the issues around current visiting policy.

ELIGIBILITY:
Arm 1

Inclusion Criteria:

* Length of stay within critical care > 4 days
* Age > 18 years
* Patients who have been admitted:

  * Following cardiac or thoracic surgery or,
  * For treatment of advanced heart failure

Exclusion Criteria:

* Pregnancy
* Diagnosed learning disability
* Pre-admission evidence of cognitive impairment
* Patients admitted to the ICU following ear nose and throat (ENT) procedures
* Patients admitted to the ICU following orthopaedics procedure
* Patients admitted to the ICU following general surgical procedures
* Patients admitted following out of hospital cardiac arrest
* Patients admitted for COVID-19 pneumonia

Arm 2

Inclusion Criteria:

For Patients:

* Length of stay within critical care > 4 days
* Age > 18 years
* Reason for admission

  * Post-operative patients following cardiac or thoracic surgery or,
  * Following admission for advanced heart failure therapies
* Provision of informed consent

For relatives:

* Age > 18 years
* Relative of a patient that has been in critical care > 4 days
* Relative of a patient who has been admitted:

  * Following cardiac or thoracic surgery or,
  * Treatment of advanced heart failure
* Relative of a patient admitted for > 4days

For Staff:

* Age > 18
* Clinical responsibility within the critical care department

Exclusion:

For patients:

* Prisoners
* Age < 18yrs
* No family or social support
* Non-English speaker
* Pre-admission evidence of cognitive impairment
* Pre-admission diagnosis of learning disability
* Imminent death
* Brain injury
* Lacks capacity (using Montreal Cognitive Assessment tool (MoCA))
* Patients admitted after out of hospital cardiac arrest
* Patients admitted to the ICU following ENT procedures
* Patients admitted to the ICU following orthopaedics procedure
* Patients admitted to the ICU following general surgical procedures
* Patients admitted with COVID-19 pneumonia

For relatives:

* Prisoner
* Age < 18yrs
* Non-English speaker
* Relative of a patient who is close to death
* Relative of a patient admitted after out of hospital cardiac arrest
* Relative of a patient admitted for ENT procedure
* Relative of a patient admitted for orthopaedic procedure
* Relative of a patient admitted following general surgical procedure

For Staff:

• Age < 18yrs

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The patient population of this unit comprises of adults undergoing cardiac or thoracic surgical procedures, the majority of which are elective operations. Other patients who receive care on this unit routinely are patients requiring level 3 care following out of hospital cardiac arrest or requiring therapies for advanced heart failure.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Duration of delirium | From the date of admission to the Intensive Care Unit (ICU) until discharge from the ICU or death, whichever came first, up to 12 months.
  Number of days patient found to have delirium using the Confusion Assessment Method for the ICU (CAM-ICU)

SECONDARY OUTCOMES:
Incidence of delirium | From the date of admission to the Intensive Care Unit (ICU) until discharge from the ICU or death, whichever came first, up to 12 months.
  CAM-ICU
Length of critical care stay | From the date of admission to the ICU until discharge from the ICU or death, whichever came first, up to 12 months.
  Days
Length of hospital stay | From the date of admission to the hospital until discharge from the hospital or death, whichever came first, up to 12 months.
  Days
Doses of specified drugs during ICU admission | From the date of admission to the ICU until discharge from the ICU or death, whichever came first, up to 12 months.
Length of time ventilated | From the date of admission to the ICU until discharge from the ICU or death, whichever came first, up to 12 months.
  Days
Mortality | 6 months

OTHER OUTCOMES:
Exploring the experiences of patients, relatives and staff of the visitation restrictions during the COVID-19 pandemic | 18 months
  Semi structured interviews

CONTACTS AND LOCATIONS:
Overall Officials: Ben Shelley, Study Chair — National Waiting Times Centre Board; Leah Hughes, Principal Investigator — National Waiting Times Centre Board

IPD SHARING:
Plan to Share IPD: Yes
Results to be published in a peer reviewed journal